CLINICAL TRIAL: NCT00965991
Title: A Randomized Prospective Trial of Metformin Compared to Glyburide in Gestational Diabetes
Brief Title: Metformin Compared to Glyburide in Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRRC#03-277
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Results first posted 2023-12-21 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; Metformin; Glyburide; oral agents
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Glyburide; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: metformin
- Glyburide (Active Comparator)
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: metformin — patients received glyburide initial dose of 500 mg PO BID. Increased as necessary to a maximum dose of 2000 mg QD to control blood glucose
  Other Names: Glucophage
  Arms: Metformin
Drug: Glyburide — Initial dose of 2.5mg PO BID increased as necessary to a maximum dose of 20 mg (10mg BID) QD to control blood glucose
  Other Names: sulfonylurea
  Arms: Glyburide

SUMMARY:
Our hypothesis is that metformin and glyburide will have equal efficacy in controlling blood glucose in gestational diabetics with no increase in adverse maternal, fetal or neonatal outcomes.

DETAILED DESCRIPTION:
Pregnant women are screened with a one hour 50g glucose challenge. Women with values of 130 mg/dl or greater are then given a 100g glucose tolerance test. Two abnormal values are diagnostic of gestational diabetes. all women are initially counseled on diet and exercise. Women who fail to maintain a fasting of <105mg/dl and 2 hr postprandial < 120 mg/dl are offered participation in the study. Women were randomized to either metformin or glyburide via a computer generated randomization. Women who fail to meet glycemic goals after receiving the maximum dose of study medication were considered treatment failures and insulin therapy was initiated.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes not controlled with diet and exercise

Exclusion Criteria:

* history of alcohol misuse
* history of drug misuse
* Chronic hypertension requiring medication
* Renal failure
* Hepatic disease or dysfunction
* Known fetal anomaly
* Inability to give consent
* known allergy to metformin or glyburide

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2023-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Moore, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Diabetes in Pregnancy Clinic, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Moore LE, Clokey D, Rappaport VJ, Curet LB. Metformin compared with glyburide in gestational diabetes: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):55-59. doi: 10.1097/AOG.0b013e3181c52132. PMID 20027034

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM 1: Metformin: Patients received metformin initial dose of 500 mg PO BID. Increased as necessary to a maximum dose of 2000 mg QD to control blood glucose
- ARM 2: Glyburide: Patients received glyburide initial dose of 2.5mg PO BID. Increased as necessary to a maximum dose of 20 mg/d to control blood glucose
Period: Overall Study
Arm/Group | ARM 1: Metformin | ARM 2: Glyburide
Started | 75 | 74
Completed | 75 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARM 1: Metformin: Metformin: Patients received glyburide initial dose of 500 mg PO BID. Increased as necessary to a maximum dose of 2000 mg QD to control blood glucose
- ARM 2: Glyburide: Glyburide: Patients received glyburide initial dose of 2.5mg PO BID. Increased as necessary to a maximum dose of 20 mg/d to control blood glucose
- Total: Total of all reporting groups
Arm/Group | ARM 1: Metformin | ARM 2: Glyburide | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 74 | 149
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7.1) | 30 (7.8) | 30 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 74 | 149

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Glucose Control
Description: The importance of exercise in the management of blood glucose was emphasized, and 30 minutes of walking per day was recommended. Patients received instruction from a nurse educator or a certified diabetes educator regarding diet and the use of the glucometer. Number of participants with a glucose level <100 mg/dL.
Time Frame: fasting and 2 hour postprandial blood glucose
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Glyburide
Number analyzed (Participants) | 75 | 74
Participants | 50 | 50

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | ARM 1: Metformin | ARM 2: Glyburide
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 0/75 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes